CLINICAL TRIAL: NCT02404467
Title: Feasibility And Safety of Early Discharge After Transfemoral Transcatheter Aortic Valve Implantation The FAST-TAVI Study
Brief Title: Feasibility And Safety of Early Discharge After Transfemoral Transcatheter Aortic Valve Implantation
Acronym: FAST-TAVI
Status: Completed | Type: Observational
Sponsor: Institut für Pharmakologie und Präventive Medizin (Network)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: FAST-TAVI
Record Dates: First submitted 2015-03-23; First posted 2015-03-31 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients receiving transfermoral TAVI: TF TAVI
  Interventions: Device: TF TAVI

INTERVENTIONS:
Device: TF TAVI — Follow-up Observation of patients having received a TF-TAVI

SUMMARY:
The hypothesis behind this study is that there is a proportion of patients considered high or intermediate risk for surgery, but relatively low risk for TAVI, which can be discharged early after the procedure (within the first 2-3 days) without additional risks. Therefore, when performed in safety, an early discharge may cut periprocedural TAVI costs significantly.

DETAILED DESCRIPTION:
TAVI (Transcatheter aortic valve Implantation) - A viable alternative to surgical aortic valve replacement for patients with severe symptomatic aortic stenosis.

Considered as being at unacceptable surgical risk. Despite its widespread utilization, there are procedure specific complications and hospitalization associated costs that limit TAVI expansion into patient populations with lower risk.

Cost-effectiveness of TAVI has been investigated either compared with standard therapy for patients who are not candidates for surgical valve replacement or with conventional surgical replacement in high-risk patients.

Formal economic evaluation in inoperable patients demonstrated that the benefits of TAVI were achieved at an acceptable incremental cost to society, at least in the context of the U.S. and U.K. health systems.

In patients with severe, symptomatic AS who are at high but not prohibitive surgical risk, the PARTNER A trial demonstrated that TAVI appeared to be an economically attractive strategy compared with aortic valve replacement, provided that patients are suitable for a transfemoral approach. On the other hand, results for trans-apical TAVI compared with surgical replacement were economically unfavorable.

ELIGIBILITY:
Inclusion Criteria:

* None

Exclusion Criteria:

* None
* Beyond the applicable criteria of the IFU no further in- and exclusion criteria are defined.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 500 consecutive patients with severe aortic stenosis selected for TF TAVI at the respective site will be enrolled. Beyond the applicable criteria of the IFU no further in- and exclusion criteria are defined.
Sampling Method: Non-Probability Sample
Enrollment: 502 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Feasibility and safety of early discharge after transfemoral (TF) TAVI (cumulative incidence of death, hospitalization, complications) | 30 days after intervention
  Cumulative incidence of a combination of all cause death, vascular Access related complications permanent Pacemaker Implantation, re-hospitalization due to cardiac reasons, and Major bleeding complications from day 4 to 30 after TAVI.

SECONDARY OUTCOMES:
Stratified Analysis of the cumulative incidence of a combination of the Primary outcome measures according to Patient risk factors and discharge date | 30 days after intervention
  Cumulative incidence of a combination of the primary outcome from day 4 to 30 in the LR / LD, HR / ED and HR / LD strata. Cumulative incidence of a combination of the primary outcome from day 4 to 15 in all strata.
Length-of-Stay after TAVI in days | 1 year
Relative costs of TAVI including hospitalization in either stratum compared to the LR / ED group | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Corrado Tamburino, MD, Principal Investigator — Ferrarotto Hospital, University of Catania; Marco Barbanti, MD, Principal Investigator — Ferrarotto Hospital, University of Catania
Locations (10):
- Italy (5):
  - Montevergine Clinic, Mercogliano, AV
  - Ferrarotto Hospital, University of Catania, Catania, Sicily
  - Universita degli studi di Bari Aldo Moro, Bari
  - University Hospital of Bologna, Policlinico S. Orsola-Malpighi (Pad.23), Bologna
  - Clinica San Gaudenzio di Novara, Novara
- Netherlands (2):
  - AMC - Academic Medical Center - University of Amsterdam, Amsterdam, AZ
  - LUMC - Leiden University Medical Center, Leiden
- United Kingdom (3):
  - Royal Vicotria Hospital, Belfast Trust, Belfast
  - Papworth Hospital, Cambridge
  - James Cook Hospital, Middlesbrough

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barbanti M, Baan J, Spence MS, Iacovelli F, Martinelli GL, Saia F, Bortone AS, van der Kley F, Muir DF, Densem CG, Vis M, van Mourik MS, Seilerova L, Luske CM, Bramlage P, Tamburino C. Feasibility and safety of early discharge after transfemoral transcatheter aortic valve implantation - rationale and design of the FAST-TAVI registry. BMC Cardiovasc Disord. 2017 Oct 10;17(1):259. doi: 10.1186/s12872-017-0693-0. PMID 29017461
- [Result] Barbanti M, van Mourik MS, Spence MS, Iacovelli F, Martinelli GL, Muir DF, Saia F, Bortone AS, Densem CG, van der Kley F, Bramlage P, Vis M, Tamburino C. Optimising patient discharge management after transfemoral transcatheter aortic valve implantation: the multicentre European FAST-TAVI trial. EuroIntervention. 2019 Jun 20;15(2):147-154. doi: 10.4244/EIJ-D-18-01197. PMID 30777842
- [Result] Spence MS, Baan J, Iacovelli F, Martinelli GL, Muir DF, Saia F, Bortone AS, Densem CG, Owens CG, van der Kley F, Vis M, van Mourik MS, Costa G, Sykorova L, Luske CM, Deutsch C, Kurucova J, Thoenes M, Bramlage P, Tamburino C, Barbanti M. Prespecified Risk Criteria Facilitate Adequate Discharge and Long-Term Outcomes After Transfemoral Transcatheter Aortic Valve Implantation. J Am Heart Assoc. 2020 Aug 4;9(15):e016990. doi: 10.1161/JAHA.120.016990. Epub 2020 Jul 25. PMID 32715844
- See also: registry on-line eCRF website — https://fast-tavi.s4trials-europe.net